CLINICAL TRIAL: NCT01488851
Title: Prospective Observational Multi Central Cohort Study to Assess the Incidence of Osteo Necrosis of Jaw in Patients With Bone Metastasis Starting Zoledronic Acid Treatment
Brief Title: Study to Assess Incidence of ONJ in Pts With Bone Mets Starting Zoledronic Acid Treatment
Status: Completed | Type: Observational
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2111-094
Record Dates: First submitted 2011-12-07; First posted 2011-12-08 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2016-01

CONDITIONS: Cancer
Keywords: Osteo necrosis of the Jaw
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prospective observational multi central cohort study to assess the incidence of osteo necrosis of jaw in cancer patient with bone metastasis starting Zoledronic acid treatment

DETAILED DESCRIPTION:
Prospective observational multi central cohort study to assess the incidence of osteo necrosis of jaw (ONJ) in pts with bone metastasis starting Zoledronic acid treatment

ELIGIBILITY:
Inclusion Criteria:

1. Bone metastasis from multiple myeloma, solid tumors, or other malignancy for which intravenous bisphosphonate has clinical indications in the treatment of metastatic bone disease.
2. All participants must be planning to receive zoledronic acid (as their sole bisphosphonate therapy) within 30 days after registration. Patients previously treated with bisphosphonate therapy are eligible if the following criteria apply:

   1. Patients may have previously received at most 3 doses of intravenous bisphosphonate therapy with ibandronate, pamidronate or zoledronic acid for low bone mass (osteopenia or osteoporosis) within 3 years prior to registration or
   2. Patients may have received intravenous bisphosphonate therapy with ibandronate, pamidronate or zoledronic acid to treat metastatic bone disease within 90 days prior to registration. Patients receiving any of these regimens for metastatic bone disease prior to 90 days before registration are not eligible, or c. Prior oral bisphosphonate therapy at any time prior to registration is allowed.
3. No pre-existing diagnosis of ONJ.
4. No history of radiation to the maxillofacial area administered for therapeutic intent in the treatment of cancer.
5. Zubrod performance status of 0-3.
6. Willing and physically able to comply with the study procedures and assessments.
7. Can concurrently participate in other therapeutic and non-therapeutic clinical trials.
8. No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.
9. Must be informed of the investigational nature of this study and must sign and give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bone Metastases
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walid Rasheed, MD, Principal Investigator — Oncology Centre, KFSH&RC
Locations (1):
- King Faisal Specialist Hospital& Research Center, Riyadh, Saudi Arabia